CLINICAL TRIAL: NCT03123276
Title: A Phase I Study to Assess the Safety and Tolerability of Pembrolizumab in Combination With Fixed Rate Gemcitabine Chemotherapy in Patients With Leiomyosarcoma and Undifferentiated Pleomorphic Sarcoma
Brief Title: Pembrolizumab and Gemcitabine Chemotherapy in Leiomyosarcoma and Undifferentiated Pleomorphic Sarcoma
Acronym: GEMMK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR 4541
Record Dates: First submitted 2017-03-31; First posted 2017-04-21 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- gemcitabine + pembrolizumab (Experimental): First cohort of 6 patients may receive Gemcitabine 800 mg/m2 + Pembrolizumab 200 mg. After safety data review, if no DLTs then dose for Gemcitabine will be increased to 1000 and further 1200 mg/m2.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — humanized IgG4 PD-1 blocking antibody
  Other Names: Keytruda
Drug: Gemcitabine — Doses of 800, 1000 and 1200 mg/m2 will be used in dose escalation phase.

SUMMARY:
Soft tissue sarcomas (STS) are a group of rare mesenchymal neoplasms affecting all ages. STS most commonly present as localised disease but despite surgery and adjuvant treatment more than half of patients will develop recurrent or metastatic disease. Leiomyosarcoma (LMS), a malignancy of smooth muscle, is one of the most common STS and undifferentiated pleomorphic sarcoma (UPS) is a common sarcoma sub-type with aggressive symptoms.

Recent studies have demonstrated reasonable sensitivity of LMS to gemcitabine monotherapy with an objective response rate of 8-19%. However the overall survival is still only about 12 months which illustrates the critical clinical need for improved therapies for advanced STS and sarcoma in general.

In this study the investigators propose to combine the immune synapse checkpoint inhibitor with the cytotoxic and immune modulating agent, gemcitabine. It is hoped that this dual immunomodulatory approach will enhance the effect of pembrolizumab on PD-L1 expressing LMS and UPS, leading to a safe treatment with patient outcomes. This is a two part, phase I, single centre dose escalation and dose expansion study in the total of 24 patients with newly diagnosed metastatic or inoperable LMS and UPS. There will be approximately 12 patients in the dose escalation cohort (part A) and the starting dose will be a fixed dose rate (FDR) gemcitabine of 800 mg/m2 on day 1 and 8 of 21 days cycles in combination of 200 mg of pembrolizumab given as an infusion on day 1 every 3 weeks. The MTD cohort (part B) will then be expanded to a total of 12 patients in order to further evaluate the safety and tolerability of that dose as well as to preliminarily assess response to therapy.

The study is sponsored by Royal Marsden NHS Foundation trust and the funding for the study is provided by Merck Sharp & Dohme Limited.

DETAILED DESCRIPTION:
This is a two part, phase I, single centre dose escalation and dose expansion study to establish the safety, tolerability and pharmacokinetics of pembrolizumab in combination with different dose levels of fixed dose rate gemcitabine in patients with newly diagnosed metastatic or inoperable leiomyosarcoma and undifferentiated pleomorphic sarcoma (UPS), for whom gemcitabine monotherapy is deemed appropriate, or in patients with previously treated leiomyosarcoma and undifferentiated pleomorphic sarcoma, not including gemcitabine, with disease progression documented in the 12 weeks prior to enrolment.

There will be a maximum of 18 patients in the dose-escalation cohort (part A) and the starting dose will be a fixed dose rate (FDR) gemcitabine of 800 mg/m2 on day 1 and 8 of 21 days cycles in combination of 200 mg of pembrolizumab given as an infusion on day 1 every 3 weeks. There will be a minimum of three and a maximum of six evaluable patients entered per dose cohort and each patient will continue to receive treatment cycles of gemcitabine in combination with pembrolizumab for as long as he/she is, in the opinion of the investigator, deriving clinical benefit and continues to meet re-treatment criteria. Treatment will continue until disease progression or is stopped because of toxicity. There will be an option to continue pembrolizumab alone in patients with SD or response who stop gemcitabine for toxicity before completing 6 cycles of combination therapy. During the dose-escalation phase, safety, tolerability, biological and clinical activity will be assessed and the maximum tolerated dose (MTD) will be established.

The MTD cohort (part B) will then be expanded to a total of 12 patients in order to further evaluate the safety and tolerability of that dose as well as to preliminarily assess response to therapy.

A mandatory tumour biopsy will be collected prior to the start of treatment for pre-treatment testing for PD-L1 expression, Immunophenotyping and extent and localization of tumour infiltrating lymphocytes and following 3 cycles of therapy for analysis of potential markers of tumour response on post-treatment tissue. Additional mandatory bloods will be collected for analysis of potential circulating immune markers. Patient genetic material will also be collected for analysis of potential markers of tumour response and future pharmacogenetic analyses. Provision of genetic material is not mandatory for participation in the main study.

Part A: Dose escalation cohort

Part A will be the dose escalation phase. Gemcitabine doses will be escalated (or de-escalated) until the non-tolerated dose (NTD) is attained and a maximum tolerated dose (MTD) is defined. A maximum of 18 patients will be recruited in cohorts of 3 to 6 patients as part of a toxicity rule-based 3+3 design. The total number of patients will depend upon the number of dose escalations and toxicities observed.

The starting dose (dose level 1) will be 800 mg/m2 of FDR gemcitabine given by 120 min IV infusion on Day 1 and Day 8 of each 3 week cycle (see Rationale for choice of starting doses). Pembrolizumab will be administered as a 200 mg IV infusion on Day 1 following the infusion of FDR gemcitabine. Pembrolizumab infusions will be repeated every 3 weeks. Each dose escalation cohort will consist of a minimum of three and a maximum of six patients.

A dose-limiting toxicity is defined as:

* Neutropenia <0.5 x 109/L for >5 days . This must be confirmed with repeat blood tests at the Royal Marsden Hospital within 6 days of the diagnosis of neutropenia.
* Febrile neutropaenia as per definition by ESMO (>38.3°C or two consecutive readings of >38.0°C for 2 hours and an absolute neutrophil count (ANC) of <0.5 x 109/L or expected to fall below <0.5 x 109/L)
* Thrombocytopenia <25 x 109/L.
* Any non-haematological CTCAE Grade 3 or 4 toxicity that is, in the opinion of the investigator, clinically significant.

The toxicities listed above must be, in the investigator's opinion, likely to be causally linked with the administration of Gemcitabine.

In the unlikely event that dose-limiting toxicity (DLT) occurs at the proposed starting dose and that dose is deemed intolerable, a second cohort of patients will be recruited and a dose of 600 mg/m2 (dose level -1). If no dose limiting toxicity (DLT) is documented, the FDR gemcitabine dose will be escalated to 1000 mg/m2 and subsequently to 1200 mg/m2 unless 2 or more patients in a single cohort have experienced DLT.

If the first patient does not experience dose-limiting toxicity by Day 14 of the first treatment cycle, two additional patients may be entered. Three patients must complete one full cycle of treatment (to day 21 of cycle 1) for a dose-escalation decision to be made.

If one of the first three patients in a cohort experiences a DLT during the first cycle, the cohort will be expanded to six patients. If 2/3 or 2/6 patients in a cohort experience DLT during the first cycle, that dose will be considered intolerable, no further dose-escalations will occur and cohort expansion of the next lowest dose (the presumed maximum tolerated dose - MTD) will commence. Only toxicities occurring during the first treatment cycle will be taken in to account for dose escalation decisions.

If a patient withdraws or is withdrawn for reasons other than DLT prior to completing Cycle 1, the patient will be replaced.

Part B: Maximum tolerated dose cohort

A total of 12 additional patients will be recruited and dosed at the MTD identified in Part A in order to ensure the tolerability and biological activity of gemcitabine in combination with pembrolizumab as well to preliminarily assess response to therapy.

Evaluation of tumour response will be according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumours) criteria. The RECIST v1.1 guidelines for measurable, non-measurable, target and non-target lesions and the objective tumour response criteria (complete response, partial response, stable disease or progression of disease) are presented in the Appendix.

All patients will have imaging performed at the end of the 3rd and the 6th cycle. After cycle 6, RECIST evaluation will be performed at the end of every third cycle for the duration of the entire study, or more frequently if it deemed necessary by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed case of undifferentiated pleomorphic sarcoma or leiomyosarcoma and be willing to consent for archival tumour material to be requested for transfer to The Royal Marsden for future review.
2. Have biopsiable disease and be willing to agree to a biopsy in order to permit acquisition of mandatory paired tumour biopsies done during screening and following 9 weeks of treatment for analysis of immunomodulation.
3. Be willing and able to provide written informed consent/assent for the trial.
4. Be over 18 years of age on day of signing informed consent.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Have measurable disease based on RECIST 1.1.
7. Have a life expectancy of >12 weeks
8. Demonstrate adequate organ function as defined in the protocol, all screening labs should be performed within 28 days of treatment initiation.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 6 months after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 6 months after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of gemcitabine that can be safely combined with pembrolizumab in the absence of dose limiting toxicities. | completion of 1 full cycle of treatment (21 days)
  primary outcome

SECONDARY OUTCOMES:
Immunophenotyping of biopsies (FFPE samples, density and phenotype of tumour infiltrating lymphocytes; CD3+, CD8+, CD45, FoxP3 and PD1) | Pre and post-treatment (9 weeks after end of treatment)
  Secondary outcome
Location of tumour infiltrating lymphocytes (proximity to tumour cells and location relative to the microvasculature; Prototype analysis software at ICR) | Up to 18 months from the first dose administered
  Secondary outcome
Response stratification according to tumour PD-L1 expression | 6 and 12 months
  Secondary outcome
preliminary evaluation of response by using RECIST v1.1 | 2 months after the last dose
  Secondary outcome

OTHER OUTCOMES:
Identify bio-markers and correlate with clinical benefit, as defined by RECIST v1.1 | Up to 18 months from the first dose administered
  Exploratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Robin Jones, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No